CLINICAL TRIAL: NCT00548639
Title: The STATIN CHOICE Decision Aid for Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-1415; ISRCTN12345678; NCI-793-0115D
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin Choice (Experimental): Statin Choice Decision Aid The provider will introduce the patient to the choice of statins using the decision aid. The patient may make a choice then or defer this choice; in all cases, the patient goes home with the Statin Choice decision aid and pamphlet.
  Interventions: Other: Statin Choice Decision Aid
- Usual Care (Sham Comparator): Control Pamphlet the provider meets with the patient to discuss treatment options in the usual fashion.
  Interventions: Other: Control Pamphlet

INTERVENTIONS:
Other: Statin Choice Decision Aid — Paper based instrument with pictures indicating level of risk.
  Arms: Statin Choice
Other: Control Pamphlet — ADA Diabetes Sheet
  Arms: Usual Care

SUMMARY:
Diabetes is a growing epidemic within the United States that disproportionately affects economically disadvantaged communities like East Harlem. As diabetic patients are at very high risk for heart disease, experts recommend an aggressive approach towards using statins in people with diabetes. However, statins and other helpful drugs are only effective if patients decide to take them. Adherence to this medication is notoriously poor and is aggravated by its required life-long use. This study is designed to test the effectiveness of a new decision aid in helping diverse, inner-city patients with diabetes understand the risks and benefits in taking statins and whether this enhanced decision making process improves their adherence to the medication.

DETAILED DESCRIPTION:
To compare the efficacy of usual consultations with or without the decision aid STATIN CHOICE in type 2 diabetic patients using or considering using statins to lower CV risk in terms of statin use, adherence, knowledge, beliefs and decisional conflict. The study team's primary hypothesis is that 3 months after the index discussion, significantly more patients randomized to STATIN CHOICE are using statins, are adherent to statins, are knowledgeable about the statin choice, and are satisfied with their decision than patients randomized to usual care consultation, and that these benefits will be achieved without deterioration in quality of life.

ELIGIBILITY:
Inclusion Criteria:

Eligible providers are

* Internists and nurse practitioners
* Provide care for patients with type 2 diabetes
* Do not plan to relocate outside the practice in the next 6 months.

Eligible patients

* Have a diagnosis of type 2 diabetes mellitus > 1 month confirmed by provider or the medical chart
* Do not take statins, but their providers identify them as eligible for this medication
* Are currently taking statins

Exclusion Criteria:

Ineligible patients

* Have, in the providers' judgment, major barriers such as hearing impairment or dementia that would compromise their participation in shared decisionmaking;
* are not available for follow-up 3 months after randomization
* are pregnant
* are under age 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Morisky medication adherence scale | 3 months
Morisky medication adherence scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States